CLINICAL TRIAL: NCT06569992
Title: Comparison of the Relationship Between Etiology and Hemodynamic Instability in Brain Death: VIS and TIES
Brief Title: Etiology and Hemodynamic Instability in Brain Death
Status: Completed | Type: Observational
Sponsor: Antalya Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Nilgun Kavrut Ozturk, Professor MD, Antalya Training and Research Hospital
Other Study IDs: 2024-CeylanM.Braindeath
Record Dates: First submitted 2024-08-20; First posted 2024-08-26 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Brain Death
Keywords: Brain death; VIS; TIES
MeSH Terms: conditions — Brain Death

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1: Spontaneous subarachnoid hemorrhage and spontaneous intracerebral hemorrhage
  Interventions: Other: VIS, TIES
- Group 2: Traumatic intracranial hemorrhage
  Interventions: Other: VIS, TIES
- Group 3: Ischemic cerebrovascular events and hypoxic-ischemic brain injury (including cases of cardiac arrest, drowning, carbon monoxide poisoning, etc.)
  Interventions: Other: VIS, TIES

INTERVENTIONS:
Other: VIS, TIES — The vasopressor and inotropic drug dosages administered during the follow-up of these patients will be recorded, and the Vasoactive-Inotropic Score (VIS) and Total Inotrope Exposure Score (TIES) will be calculated.

SUMMARY:
Brain death is a complex and irreversible condition marked by the cessation of all brain activity. This retrospective study analyzes ICU patients who progressed from initial brain injury to brain death. The research focuses on demographic profiles, pharmacological interventions, laboratory data, and imaging findings to understand these cases clinical trajectories and therapeutic responses. Central to this study is evaluating cardiovascular support using the Vasoactive-Inotropic Score (VIS) and Total Inotrope Exposure (TIE) Score. This study explores the relationship between the etiology of brain death and the pharmacologic cardiovascular support administered, as quantified by VIS and TIES scores. This study seeks to enhance the management strategies and improve outcomes for patients diagnosed with brain death

DETAILED DESCRIPTION:
This study undertakes a comprehensive retrospective analysis of patients admitted to the intensive care unit (ICU) with an initial diagnosis of brain injury who subsequently progressed to brain death. The investigation will meticulously assess these patients, demographic profiles, pharmacological interventions, laboratory parameters, and radiological imaging findings. The overarching aim is to delineate the clinical trajectory and therapeutic responses of patients diagnosed with brain death, critically evaluating the complexities encountered during their management, and providing evidence-based insights to inform future treatment protocols.

Central to this study is the quantitative assessment of hemodynamic stability using the Vasoactive-Inotropic Score (VIS) and the Total Inotrope Exposure (TIE) Score. The VIS will quantify the need for vasopressor and inotropic support, reflecting the severity of cardiovascular instability. At the same time, the TIE Score will measure the cumulative exposure to inotropic agents, providing a comprehensive evaluation of the overall cardiovascular burden. The primary aim of this study is to explore the relationship between the etiology of brain death and the pharmacologic cardiovascular support administered, as quantified by VIS and TIES scores. Additionally, the study will assess how these pharmacologic interventions differ in patients who have undergone decompressive surgery compared to those who have not.

This thesis aspires to make a significant contribution to the optimization of management strategies for patients diagnosed with brain death, aiming to enhance clinical decision-making and improve patient outcomes in this critically ill cohort.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years) admitted to the intensive care unit (ICU) at Antalya Training and Research Hospital between 2019 and 2023.
* Patients with a confirmed diagnosis of brain death based on a positive apnea test and/or neuroimaging findings.
* Patients with comprehensive and complete clinical data available in the hospital's medical records.

Exclusion Criteria:

* Patients under the age of 18.
* Patients with incomplete clinical data in the medical records.
* Patients with moderate to severe heart failure.
* Patients with major organ injuries in addition to traumatic intracranial hemorrhage.
* Pregnant patients.
* Patients with significant comorbidities that could impact hemodynamic stability.
* Patients experiencing hemodynamic instability due to septic shock.
* Patients who were initially treated for brain injury at external facilities and later transferred to our hospital.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will retrospectively analyze data from patients diagnosed with brain death and followed in the Anesthesiology and Intensive Care Units at University of Health Science Antalya Training and Research Hospital between January 1, 2019, and December 31, 2023. Patients will be categorized based on the etiological cause of brain injury into the following groups: those with spontaneous subarachnoid hemorrhage and spontaneous intracerebral hemorrhage (Group 1), those with traumatic intracranial hemorrhage (Group 2), and those with ischemic cerebrovascular events and hypoxic-ischemic brain injury (including cases of cardiac arrest, drowning, carbon monoxide poisoning, etc.) (Group 3).
Sampling Method: Non-Probability Sample
Enrollment: 216 (Actual)
Dates: Start 2024-05-30 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Total Inotrope Exposure Score (TIES) | From beginning to vasoactive-inotropic drugs infusion until diagnosis of brain death, 10 days (with intermediate measurements every hours)
  Dopamine dose (μg/kg/min) × [length of administration in days] + Dobutamine dose (μg/kg/min) × [length of administration in days] + 10 × Milrinone dose (μg/kg/min) × [length of administration in days] + 100 × Epinephrine dose (μg/kg/min) × [length of administration in days] + 100 × Norepinephrine dose (μg/kg/min) × [length of administration in days] + 10,000 × Vasopressin dose (U/kg/min) × [length of administration in days
Vasoactive-Inotropic Score (VIS) | From beginning to vasoactive-inotropic drugs infusion until diagnosis of brain death, 10 days (with intermediate measurements every hours)
  Dopamine dose (μg/kg/min) + dobutamine dose (μg/kg/min) + 100 × epinephrine dose (μg/kg/min) + 10 × milrinone dose (μg/kg/min) + 10 000 × vasopressin dose (unit/kg/min) + 100 × norepinephrine dose (μg/kg/min).

CONTACTS AND LOCATIONS:
Overall Officials: Nilgun Kavrut Ozturk, Professor, Study Chair — University of Health Science Antalya Training and Research Hospital
Locations (1):
- University of Health Sciences, Antalya, Muratpasa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Flowers WM Jr, Patel BR. Persistence of cerebral blood flow after brain death. South Med J. 2000 Apr;93(4):364-70. PMID 10798503
- [Result] Belletti A, Lerose CC, Zangrillo A, Landoni G. Vasoactive-Inotropic Score: Evolution, Clinical Utility, and Pitfalls. J Cardiothorac Vasc Anesth. 2021 Oct;35(10):3067-3077. doi: 10.1053/j.jvca.2020.09.117. Epub 2020 Sep 22. PMID 33069558